CLINICAL TRIAL: NCT06798961
Title: Longitudinal Evaluation of Active-Duty Personnel with Accessory Pathways (LEAD-AP)
Acronym: LEAD-AP
Status: Active, not recruiting | Type: Observational
Sponsor: United States Naval Medical Center, San Diego (U.S. Federal Agency)
Responsible Party: Principal Investigator, Abiola Babawale, Principal Investigator, United States Naval Medical Center, San Diego
Other Study IDs: NMCSD.2024.0019
Record Dates: First submitted 2025-01-23; First posted 2025-01-29 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-01

CONDITIONS: Cardiac Death; Cardiac Death, Sudden; Wolf Parkinson White Syndrome
Keywords: accessory pathway; ablation; cardiac death; Wolf Parkinson's white
MeSH Terms: conditions — Death; Death, Sudden, Cardiac; Wolff-Parkinson-White Syndrome; Pre-Excitation Syndromes | interventions — Standard of Care

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- All patients: Patients diagnosed with Accessory pathway between ages 18-40.
  Interventions: Procedure: Ablation; Procedure: Standard of care without ablation

INTERVENTIONS:
Procedure: Ablation — Patient treated with an ablation to eliminate the accessory conduction pathway in the heart.
Procedure: Standard of care without ablation — Patient diagnosed with accessory pathway but elected against cardiac ablation as a treatment option at the time of diagnosis.

SUMMARY:
The investigators propose a secondary chart review using EMR data to identify risk factors for sudden cardiac death in active-duty members diagnosed with an accessory pathway between the ages of 18-40.

DETAILED DESCRIPTION:
The LEAD-AP study is a dual arm retrospective observational cohort study (using existing records) to investigate the long-term outcomes of patients diagnosed with an accessory pathway during their military service.

Overall objective: Identifying additional risk factors associated with sudden cardiac death to help with risk stratification and guide ablation criteria for patients diagnosed with accessory pathways between the ages of 18-40.

Specific Aim/Research Question: The investigators will evaluate whether patients with an ablation have improved outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Active Duty between ages 18-40 who were diagnosed with an accessory pathway between 1/1/1990 - 5/30/2024.

Exclusion Criteria:

* Patient without the diagnosis of Wolf Parkinson's White (WPW) syndrome

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Active Duty between ages 18-40 who were diagnosed with an accessory pathway between 1/1/1990 - 5/30/2024.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Cardiac death | 5 years
  The goal of LEAD AP is to investigate the long-term outcomes of patients diagnosed with an accessory pathway during their military service; with the goal of identifying additional risk factors associated with sudden cardiac death to help with risk stratification and guide ablation for patients diagnosed with accessory pathways between the ages of 18-40.

CONTACTS AND LOCATIONS:
Locations (1):
- Naval Medical Center San Diego, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Zipes DP, Link MS, Ackerman MJ, Kovacs RJ, Myerburg RJ, Estes NA 3rd; American Heart Association Electrocardiography and Arrhythmias Committee of Council on Clinical Cardiology, Council on Cardiovascular Disease in Young, Council on Cardiovascular and Stroke Nursing, Council on Functional Genomics and Translational Biology, and American College of Cardiology. Eligibility and Disqualification Recommendations for Competitive Athletes With Cardiovascular Abnormalities: Task Force 9: Arrhythmias and Conduction Defects: A Scientific Statement From the American Heart Association and American College of Cardiology. Circulation. 2015 Dec 1;132(22):e315-25. doi: 10.1161/CIR.0000000000000245. Epub 2015 Nov 2. No abstract available. PMID 26621650
- [Background] Huang SY, Hu YF, Chang SL, Lin YJ, Lo LW, Tuan TC, Lee PC, Li CH, Suenari K, Chao TF, Tai CT, Chiang CE, Chen SA. Gender differences of electrophysiologic characteristics in patients with accessory atrioventricular pathways. Heart Rhythm. 2011 Apr;8(4):571-4. doi: 10.1016/j.hrthm.2010.12.013. Epub 2010 Dec 13. PMID 21147259
- [Background] Cain N, Irving C, Webber S, Beerman L, Arora G. Natural history of Wolff-Parkinson-White syndrome diagnosed in childhood. Am J Cardiol. 2013 Oct 1;112(7):961-5. doi: 10.1016/j.amjcard.2013.05.035. Epub 2013 Jul 2. PMID 23827401
- [Background] Obeyesekere MN, Leong-Sit P, Massel D, Manlucu J, Modi S, Krahn AD, Skanes AC, Yee R, Gula LJ, Klein GJ. Risk of arrhythmia and sudden death in patients with asymptomatic preexcitation: a meta-analysis. Circulation. 2012 May 15;125(19):2308-15. doi: 10.1161/CIRCULATIONAHA.111.055350. Epub 2012 Apr 24. PMID 22532593
- [Background] Pediatric and Congenital Electrophysiology Society (PACES); Heart Rhythm Society (HRS); American College of Cardiology Foundation (ACCF); American Heart Association (AHA); American Academy of Pediatrics (AAP); Canadian Heart Rhythm Society (CHRS); Cohen MI, Triedman JK, Cannon BC, Davis AM, Drago F, Janousek J, Klein GJ, Law IH, Morady FJ, Paul T, Perry JC, Sanatani S, Tanel RE. PACES/HRS expert consensus statement on the management of the asymptomatic young patient with a Wolff-Parkinson-White (WPW, ventricular preexcitation) electrocardiographic pattern: developed in partnership between the Pediatric and Congenital Electrophysiology Society (PACES) and the Heart Rhythm Society (HRS). Endorsed by the governing bodies of PACES, HRS, the American College of Cardiology Foundation (ACCF), the American Heart Association (AHA), the American Academy of Pediatrics (AAP), and the Canadian Heart Rhythm Society (CHRS). Heart Rhythm. 2012 Jun;9(6):1006-24. doi: 10.1016/j.hrthm.2012.03.050. Epub 2012 May 10. No abstract available. PMID 22579340
- [Background] Page RL, Joglar JA, Caldwell MA, Calkins H, Conti JB, Deal BJ, Estes NA 3rd, Field ME, Goldberger ZD, Hammill SC, Indik JH, Lindsay BD, Olshansky B, Russo AM, Shen WK, Tracy CM, Al-Khatib SM; Evidence Review Committee Chairdouble dagger. 2015 ACC/AHA/HRS Guideline for the Management of Adult Patients With Supraventricular Tachycardia: A Report of the American College of Cardiology/American Heart Association Task Force on Clinical Practice Guidelines and the Heart Rhythm Society. Circulation. 2016 Apr 5;133(14):e506-74. doi: 10.1161/CIR.0000000000000311. Epub 2015 Sep 23. No abstract available. PMID 26399663